CLINICAL TRIAL: NCT01219478
Title: Research of the Correlation Between Metabolic Syndrome, Retinal Thickness and Visual Acuity
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Hui-Chun Ho, Department of Ophthalmology, Wanfang Hospital
Other Study IDs: 99028
Record Dates: First submitted 2010-10-10; First posted 2010-10-13 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-12

CONDITIONS: Visual Acuity
Keywords: To investigate the relationship between retinal thickness (RT) and metabolic risks (MRs) in patients without retinal lesion

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- control: 0 metabloil risk
- 1: 1 metabloil risk
- 2: 2 metabloil risk
- 3: 3 metabloil risk

SUMMARY:
Purpose: To investigate the relationship between retinal thickness (RT) and metabolic risks (MRs) in patients without retinal lesion.

Methods: Fifty-two patients over 60 y/o were divided into four groups according to their MRs of hypertension, hyperlipidemia or hyperglyceremia. After complete ophthalmic examination, optical coherence tomography was performed to measure RT.

ELIGIBILITY:
Inclusion Criteria:

* We enrolled the patients included age more than 60 years old, no positive finding during dilated fundus examination.

Exclusion Criteria:

* The exclusion criteria were as followed:

  * systemic disease that will affect visual acuity evaluation (for example: CVA), *opaque cornea and vitreous
  * glaucoma
  * uvietis and other clinically established ocular disease.
* According to the LOCS III11, those who had nuclear opalescence, nuclear color more than grade 3 or any grade of cortical cataract and posterior subcapsular cataract were also eliminated.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who were over 60 y/o were divided into four groups according to their MRs of hypertension, hyperlipidemia or hyperglyceremia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-01; Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chun Ho, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan